CLINICAL TRIAL: NCT01640496
Title: Vitamin D Treatment in Ulcerative Colitis
Acronym: Vitamin D
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: North Shore University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-0542
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Disease
Keywords: Ulcerative Colitis; Inflammatory Bowel disease; IBD; Vitamin D
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Active Comparator): Subjects will take 1 pill per day for 8 weeks.
  Interventions: Drug: Vitamin D3
- Placebo (Placebo Comparator): Subjects will be asked to take 1 pill per day for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — 3000 IU Vitamin D3 tablets (Cholecalciferol) will be used. 28 pills per bottle. Subjects will be given 2 bottles to be taken for the duration of this study.
  Other Names: Cholecalciferol
  Arms: Vitamin D
Other: Placebo — Placebo will be given to subjects. 28 pills per bottle. Subjects will be given 2 bottles to be taken for the duration of this study.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test blood and tissue samples of people with Ulcerative Colitis (UC) to see what effects Vitamin D3 may have on the immune system. This research is being done because it could lead to the development of new treatment for people with Inflammatory Bowel Disease (IBD).

DETAILED DESCRIPTION:
The primary endpoint of the trial is the change in colonic permeability as a global assessment of vitamin D3 effects throughout the colon in patients with Ulcerative Colitis. Secondary endpoints will be changes in colonic tight junction protein expression, and their relationship to serum vitamin D level, VDR expression, inflammatory cytokines, and histologic inflammation

ELIGIBILITY:
Inclusion Criteria:

* Patients must be over 18 years of age
* have a diagnosis of UC as confirmed by histology.
* UC patients must have active but mild disease as confirmed by a Mayo Clinic endoscopy score from 2-4,
* not requiring medication adjustment during the trial.
* Patients must be capable of understanding the purpose, risks and expectations of study participation and willing to provide written informed consent.

Exclusion Criteria:

* Individuals on vitamin D or laxative therapy (except for purposes of endoscopy preparation),
* UC patients with fulminant colitis or active C difficile or other colonic infections,
* age<18 year old,
* individuals with bleeding disorders will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Mucosal Permeability | 8 weeks
  The primary endpoint of the trial is the change in colonic permeability as a global assessment of vitamin D3 effects throughout the colon in patients with Ulcerative Colitis.

SECONDARY OUTCOMES:
Mucosal tight junction protein expression | 8 weeks
  Secondary endpoints will be changes in mucosal tight junction protein expression, and their relationship to serum vitamin D level, VDR expression, inflammatory cytokines, and histologic inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Pekow, M.D., Principal Investigator — University of Chicago
Locations (1):
- NorthShore, Evanston, Illinois, United States